CLINICAL TRIAL: NCT06865950
Title: Sex Differences in Prehospital Acute Management of Suspected Stroke Patients
Brief Title: Sex diffErences in prehoSpitAl Stroke MEdicine
Acronym: SESAME
Status: Recruiting | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Collaborators: East of England Ambulance Service NHS Trust (Other Government); Norwegian Air Ambulance Foundation (Other); Glasgow Caledonian University (Other); Assiut University (Other); The George Institute (Other); Hospital de Clinicas de Porto Alegre (Other); Hospital Israelita Albert Einstein (Other); University Of Perugia (Other); University "Ss Cyril and Methodius", North Macedonia (Unknown); 115 People's Hospital (Other Government); Selcuk University (Other); Copenhagen University Hospital, Denmark (Other); National University Hospital, Singapore (Other); Kwame Nkrumah University of Science and Technology, Ghana (Unknown); Catholic University of Health and Allied Sciences, Mwanza, Tansania (Unknown)
Responsible Party: Sponsor
Other Study IDs: SESAME_137/2024
Record Dates: First submitted 2025-01-24; First posted 2025-03-10 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-01

CONDITIONS: Stroke Acute; Emergency Medical Services; Sex Characteristics; Prehospital Setting
Keywords: stroke; sex differences; ambulance service; stroke treatment; inequality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dispatch centre suspected stroke patients: Patients with dispatch centre suspected acute stroke diagnosis, who therefore had a code stroke dispatch
- Patients with EMS on scene suspected acute stroke diagnosis: Patients for which the EMS at the emergency side suspects an acute stroke diagnosis and deliver the EMS stroke protocol treatment.
- Patients with hospital confirmed acute stroke diagnosis: Patient who received a final hospital diagnosis of stroke after full diagnostic work-up.

SUMMARY:
Background: Stroke is a leading cause for individual, family and societal harm with huge health-economic impact. Immediate and correct prehospital acute stroke pathway initiation is key for treatment success.

Evidence points towards sex inequity in management pathways of acute stroke care. A complicating factor in acute stroke management is the diversity in clinical presentation among patients of different sex. This increases the challenges of correct prehospital identification.

Most of the currently available data on male and female differences in acute stroke management come from patients with hospital-confirmed stroke. Little to no information is available about sex-related management differences of patients with prehospital suspected stroke, often missed by stroke quality databases.

Objectives: To identify sex differences in EMS-delivered prehospital diagnostic accuracy and management of patients with suspected or confirmed acute stroke.

Methods: International project collaboration to conduct a cross-regional cohort analysis of patients with a prehospital working diagnosis of stroke and/or hospital-confirmed stroke diagnosis.

Relevance: More information and details about the reasons for a potential prehospital treatment inequity are a necessary next step for any improvement and subsequent development of structured training programmes for emergency medical service personnel. This project is the first large-scaled international collaboration addressing sex differences in prehospital stroke care. With this approach the project will not only lead to more urgently needed information, but will also serve as a lighthouse project for raising general awareness for this topic.

DETAILED DESCRIPTION:
Current state of research in the field Acute stroke patients need an optimal prehospital management with rapid identification of their suspected stroke and high quality prehospital care to gain access to modern hyperacute stroke treatments. The fewer barriers there are to a fast response, the better the patient's outcome will be. However, research results indicate that women are disadvantaged in their prehospital care by often receiving wrong working diagnosis, delayed management and less structured prehospital acute stroke care.

This is nourished by the fact that Emergency Medical Service (EMS) clinicians, who are responsible for this rapid management are usually not specialised in stroke medicine, which results in reported numbers of missed stroke diagnosis of as high as 52% (Jones, Bray et al. 2021). Prehospital identification is additionally impeded by several factors, including the limited diagnostic equipment available at the emergency site, the broad variety of non-stroke diseases presenting with stroke-like symptoms (Gibson and Whiteley 2013) and not least the time pressure behind identification of stroke suspects following the "time is brain" concept. In many areas, stretched hospital emergency departments (ED) pushing towards pathways for admission avoidance, add further challenges by increasing the aim to manage as many as possible patients in the community. Especially those patients, who present as stroke-mimics to the EMS (patients with stroke like symptoms, that are not caused by a stroke) and patients with general symptoms like dizziness or confusion could be left behind under this pressure (Neves Briard, Zewude et al. 2018).

Further complicating is that not all acute stroke patients present with the classical face, arm (leg), speech abnormalities. Especially, women often show non-traditional stroke symptoms like the ubiquitous symptoms of altered mental status, headache, reduced consciousness, generally reduced condition or dizziness (Lisabeth, Brown et al. 2009, Girijala, Sohrabji et al. 2017, Bushnell, Howard et al. 2018, Carcel, Woodward et al. 2020, Patti and Gupta 2022, Shajahan, Sun et al. 2022). This makes the already challenging stroke diagnosis even more difficult.

Information available on gender inequality of prehospital and hyperacute stroke care is growing (Walter, Phillips et al. 2022). Some studies report patient-dependent delays as underlying factors for a later arrival at hospital (Mainz, Andersen et al. 2020), but more and more pieces of information point towards an additional impact of health system-caused sex inequity in prehospital stroke pathways. A drawback of many results is the analysis of hospital-confirmed stroke patient cohorts, which carry the selection bias of missing patients, who never got diagnosed as acute stroke victims (Volpe, Zuniga et al. 2023).

Sex-related inequality in prehospital assessment of stroke patients may have potentially devastating consequences. A very recent Australian population-based cohort study with more than 200,000 confirmed stroke patients with analysis of prehospital management, identified that women, especially those younger than 70 years of age, were less likely than men to receive immediate stroke assessment despite their more frequent admission to hospital by ambulance, which is known to be an important initiating factor for rapid specialist care (Wang, Carcel et al. 2022). In the same study, it could be identified that women with stroke were more often assessed for headache, anxiety and emotional distress and, therefore, did not receive prehospital stroke care according to standard EMS protocols. A Californian state-wide database analysis of >300,000 patients identified that the probability for women to get correctly identified as suspected stroke patients in the prehospital setting was 26% lower and this was likely caused by the different clinical presentations (Govindarajan, Friedman et al. 2015). No information about any resulting differences in the subsequent acute stroke treatment, like e.g. administration rates of recanalising therapies was analysed.

A systematic metanalysis of 21 observational studies with nearly 7,000 stroke patients focused on the type of symptom as a most important factor for correct prehospital diagnosis. More than a quarter of all stroke patients missed by the prehospital teams presented with non-classical symptoms (Jones, Bray et al. 2021). In a very recent study with more than 5000 acute stroke patients in Sweden, Magnusson and co-authors identified that patients correctly identified as stroke suspects in the prehospital setting less frequently had a decreased level of consciousness, which is a common non-traditional stroke symptom in women. Most importantly, they found that identification of a stroke diagnosis at the emergency site was not only associated with an earlier arrival at a stroke unit and increased rate of acute stroke recanalising treatments, but also with a lower risk of death during 3 months of follow-up (Magnusson, Herlitz et al. 2022).

Data available for hyperacute treatment access vary by country. A German nationwide cohort analysis with >1 million patients identified a higher probability of men receiving stroke unit treatment (OR, 1.11; 95% CI, 1.09-1.12) with a lower in-hospital mortality (OR, 0.91; 95% CI, 0.89-0.93) compared to women (Weber, Krogias et al. 2019). However, IVT treatment numbers were similar in this study and more women received endovascular treatment (EVT). A Swedish analysis confirmed significantly lower numbers of women receiving stroke unit care in their cohort (Dahl, Hjalmarsson et al. 2020). In contrast to the German analysis, the American Get-With-The-Guidelines-Stroke registry identified female sex as a risk factor for not receiving IVT in their retrospective cohort analysis of acute ischaemic stroke patients, arriving at hospital within 2 hours after symptom onset (Messe, Khatri et al. 2016).

Evidence addressing differences in prehospital stroke care mostly comes from single countries and cohort studies of confirmed acute stroke patients, not always focused on sex differences. Therefore, these analyses often contain a certain population selection bias, which may influence their sex-related results. So far, no multi-national analysis has been performed investigating both, prehospital and hospital-diagnosed stroke patients with regards to sex differences. Additionally, it is likely that equity in prehospital stroke treatment strongly depends on the quality of stroke education of EMS staff, and this varies between countries and regions. However, there is only scarce information available directly addressing the awareness of EMS clinicians for sex differences in stroke presentation, while this is a fundamental part of EMS education for myocardial infarcts.

Studies are needed to gain more information about the current knowledge of EMS clinicians about varying stroke symptoms and to identify differences in management not only in hospital cohorts, but also in patients with prehospital stroke diagnosis. These are first steps for change and towards the development an adjusted educational programme, which can help to tackle potential sex inequities.

Scientific relevance and socioeconomic impact of the research project Research data indicates existing management inequity in prehospital stroke care, which could carry over to in-hospital pathways and subsequent access to high quality stroke treatment. Little to no data is available which addresses sex inequities in prehospital treatment and the role EMS clinicians play in this.

This knowledge gap must be closed as women show a higher stroke incidence and prevalence than men (incidence 6.44 million to 5.79 million; prevalence 56.4 million to 45.0 million (Collaborators 2021). This implies an ethical need to understand and tackle potential inequalities. This also bears a huge socio-economic relevance. A recent meta-analysis identified costs per patient per year of up to $84,900 for e.g. haemorrhagic stroke treatment in South Korea and life time costs of up to $232,100 in Australia (Strilciuc, Grad et al. 2021), emphasising the financial relevance of optimised access to high quality stroke care to every member of the society. In addition, a recent Canadian population-based cohort analysis identified that care costs for complex continuing care, long-term care, and home care after stroke were higher in women than men, adding to the monetary burden of the disease (Yu, Krahn et al. 2021).

The traditional view that symptom presentation and treatment is the same across sex is slowing down to preventing the establishment of equity in care. As of now, no study has collected information about existing sex differences in prehospital stroke care in multiple countries combined with an analysis of existing knowledge among prehospital and emergency staff.

The proposed project would be the first multinational cohort study to address and analyse such differences in prehospital stroke pathways. Patients treated in the years 2024 and 2025 will be analyzed either retrospectively or prospectively.

ELIGIBILITY:
Inclusion Criteria:

* For all participants:
* Adults aged 18 years of age and older
* Emergency call to the national emergency telephone number because of acute symptoms
* EMS treatment

For cohort 1:

- Working diagnosis of acute stroke or TIA raised by the emergency medical dispatch centre

For cohort 2:

- Working diagnosis of acute stroke or TIA raised by the EMS personnel at the emergency site

For cohort 3:

- Hospital confirmed diagnosis of acute stroke or TIA

Exclusion Criteria:

* Patients, who have acute stroke symptoms but do not involve the EMS and make their way to hospital themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for cohorts 1 and 2 patients will be identified through information coming from the prehospital patient records. All patients with prehospital suspected diagnosis of stroke or TIA will be considered. Terminology will be adjusted to local terms.
  Cohort 3 patients will be identified in the stroke department if diagnosed with stroke (ischaemic or haemorrhagic) or TIA.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prehospital management accuracy | 36 hours after emergency call
  Proportion of patients with correct prehospital stroke management defined as correct prehospital working diagnosis compared with hospital diagnosis and adherence to local prehospital stroke guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Saarland University, Homburg, Germany

IPD SHARING:
Plan to Share IPD: No
The original data will be owned by the individually participating researchers and centres. The overall study group does not own any data, hence cannot share any individual participant information.